CLINICAL TRIAL: NCT06251115
Title: Clinical Study on the Safety and Efficacy of QY-1-T in the Treatment of HBV-associated Advanced Liver Cancer
Brief Title: Clinical Study on the Safety and Efficacy of QY-1-T in the Treatment of HBV-associated Advanced HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shenzhen Zhongke Qiyuan Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Jiang Long, Chief physician of hepatobiliary and pancreatic surgery, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-QY-1-T
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Liver Cancer
Keywords: TCR- T; HBV-HCC; Immunotherapy; Liver cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QY-1-T (Experimental): Each patient will undergo a core study of approximately 1 year after enrollment: including screening period, apheresis, first treatment cycle (induction phase), observation period, second treatment cycle (maintenance phase), and routine follow-up period.
  The first treatment cycle (induction period): It is planned to use 4 induction doses of 1×10^4 cells/Kg, 1×10^5 cells/Kg, 1×10^6 cells/Kg, 5×10^6 cells/Kg or 10×10^6 cells/Kg respectively on day 1 ( C1D1), day 8 (C1D8), day 15 (C1D15) and day 22 (C1D22) received stepped dosing of QY-1-T. A 30-day medical observation will be conducted after the first treatment cycle, followed by the second treatment cycle.
  Second treatment cycle: The dose is 5×10^6 cells/Kg or 10×10^6 cells/Kg. TCR-T was infused once a week, that is, QY-1-T administration was performed on day 1 (C2D1), day 8 (C2D8), day 15 (C2D15), and day 22 (C2D22).
  Interventions: Drug: QY-1-T

INTERVENTIONS:
Drug: QY-1-T — QY-1-T is a TCR-T drug targeting HBV-related HCC

SUMMARY:
The vast majority of liver cancers have an insidious onset and are often asymptomatic in the early stages, making early diagnosis difficult. Once diagnosed, most liver cancers have reached locally advanced stages or distant metastases, equivalent to Barcelona stage (BCLC) C-D. The tumors progress rapidly and there is a lack of effective treatments. The survival period of cancer patients is generally only 3-6 months. Cellular immunotherapy, including CAR-T and TCR-T, is considered a new hope for the treatment of cancer.

The purpose of this study is to explore the safety of QY-1-T (a TCR-T targeting HBV) in the treatment of HBV-related liver cancer, and to preliminarily evaluate the efficacy of QY-1-T in patients with HBV-related advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-75 years old (male or female)
2. The subject voluntarily participate and have the ability to sign the informed consent independently
3. Patient with advanced hepatocellular carcinoma (HCC) confirmed by histopathology or cytology (BCLC stage B and C, or CNLC stage IIA/IIB and IIIA/IIIB). One of the following four conditions applies:a. Patients with advanced hepatocellular carcinoma (HCC) who are not candidates for surgery or local therapy and have previously failed or become intolerable after at least second-line or higher standardized systemic therapy (including but not limited to targeted therapy, immunotherapy, or chemotherapy) and whose disease progression or intolerance has been determined by imaging examination during or after treatment, Or patients whom the investigator believes could benefit. b. HCC patients with clinically confirmed recurrence or progression after local treatment, and the interval between treatment and enrollment is at least 4 weeks. c. HCC recurrence after resection progresses or is not tolerated by systemic therapy or TACE/HAIC or radiofrequency ablation, and the interval between treatment and entrainment is at least 4 weeks. d. Recurrence of liver cancer after liver transplantation progresses or is not tolerated after systemic therapy or TACE/HAIC or radiofrequency ablation, and the interval between treatment and entrainment is at least 4 weeks
4. Prior systemic therapy should be discontinued for at least 2 weeks prior to enrollment
5. The expected survival time is more than 6 months
6. The subject has at least one tumor lesion that can be measured according to RECIST1.1
7. Hepatitis B virus surface antigen (HBsAg) positive or previous positive history
8. The HLA typing of peripheral blood was HLA-A*11:01
9. Non-cirrhosis or compensatory cirrhosis Child-Pugh < 7 score
10. ECOG scoring standard ≤1
11. Blood routine and blood biochemical indicators: a. white blood cells ≥3×10^9/L. b. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤5× upper limit of normal (ULN). c. Serum total bilirubin ≤2×ULN. d.eGFR≥60ml /min. e. Hemoglobin > 90g/L. f. Platelet count ≥50×10^9/L. g. Creatinine ≤1.5×ULN. h. International standardized ratio INR≤1.5 or activated partial thrombin time (APTT) extended within 10s.
12. Female subjects of childbearing age, whose serum pregnancy tests must be negative, and all subjects must agree to take effective contraceptive measures during the test
13. Subject agrees to abstain from alcohol during the study
14. The subject is willing and able to follow all treatment procedures and protocols

Exclusion Criteria:

1. The presence of a secondary primary malignancy, except in the following cases: a. Non-melanoma treated by excision, such as basal cell skin cancer. b. curable carcinoma in situ, such as cervical, bladder or breast cancer
2. Liver tumor load exceeds 70%
3. Co-transplanters
4. Main portal vein cancer thrombus
5. Moderate to severe ascites
6. Human immunodeficiency virus (HIV) 1 or 2 positive or acquired immunodeficiency syndrome (AIDS) history, treponema pallidum antibody positive
7. Decompensated cirrhosis Child-Pugh B or C (7-15 points)
8. Clinically significant bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, hereditary or acquired bleeding and thrombosis tendency (such as hemophilia, coagulation disorder, thrombocytopenia, hypersplenism, etc.) within 2 weeks prior to the study, and more serious arteriovenous thrombosis events occurring within the previous 6 months,Such as cerebrovascular diseases (including cerebral hemorrhage, cerebral infarction), pulmonary embolism, etc.
9. Have high blood pressure that cannot be effectively controlled, i.e. systolic blood pressure > 160 mmHg or diastolic blood pressure > 110 mmHg after antihypertensive treatment
10. Serum HBV DNA≥1000 IU/ml during screening (HBV positive for transplant donors of primary liver cancer patients), antiviral treatment can be performed according to the actual situation before admission
11. HCV RNA positive
12. Prior cell therapy, such as but not limited to NK, CIK, DC, CTL, stem cell therapy
13. Concurrent treatment with other anti-tumor therapies, including cytotoxic chemotherapy, hormone therapy and immunotherapy
14. Use of immune checkpoint inhibitors within 1 month
15. Patient with Grade III or IV cardiac dysfunction, arrhythmias that cannot be controlled by drugs or QTc interval > 450ms for men and > 470ms for women according to the NYHA grading criteria
16. Any other medical conditions that may increase subjects' risk or interfere with study results
17. Has any condition that interferes with drug administration and study sample collection
18. Those who have a history of psychotropic drug abuse and cannot abstain or have a history of mental disorders
19. Participate in other drug clinical studies within 4 weeks before screening
20. Pregnant or lactating women
21. Failure to follow or cooperate with relevant treatment procedures and protocols during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with adverse events (AEs) and laboratory abnormalities defined as dose limiting toxicities (DLT) | Up to 1 month after the last infusion
  To assess the tolerability of QY-1-T and determine the maximum tolerated dose (MTD)

SECONDARY OUTCOMES:
Efficacy: antitumor activity of QY-1-T in subjects with HBV-related HCC | Up to 1 year after the last infusion
  Tumor response assessment in accordance with mRECIST and iRECIST

OTHER OUTCOMES:
Efficacy: antiviral activity of QY-1-T | Up to 1 year after the last infusion
  Changes in serum levels of hepatitis B surface antigen (HBsAg) before and after QY-1-T infusion
Efficacy: antiviral activity of QY-1-T | Up to 1 year after the last infusion
  Changes in serum levels of hepatitis B virus deoxyribonucleic acid (HBV-DNA) before and after QY-1-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Long, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China